CLINICAL TRIAL: NCT07404592
Title: TRACHEOSTOMY PRACTICES IN ADULT INTENSIVE CARE UNITS IN IZMIR, TURKEY: A MULTICENTRE POINT-PREVALENCE STUDY
Brief Title: Tracheostomy Practices in Adult Intensive Care Units: A Multicentre Study in Izmir
Acronym: IZ-TRACH
Status: Completed | Type: Observational
Sponsor: Izmir City Hospital (Other Government)
Responsible Party: Principal Investigator, Murat Kaykaç, Anesthesiology and Reanimation Specialist, MD, Izmir City Hospital
Other Study IDs: 2025/352
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Tracheostomy
Keywords: Tracheostomy; Intensive care unit; Mechanical ventilation; Multidisciplinary decision-making; Point-prevalence study
MeSH Terms: interventions — Tracheostomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tracheostomy Patients: Adult patients (aged ≥18 years) hospitalized in intensive care units who have undergone either surgical or percutaneous tracheostomy.
  Interventions: Procedure: Tracheostomy

INTERVENTIONS:
Procedure: Tracheostomy — The application of surgical or percutaneous dilatational tracheostomy (Griggs guidewire dilating forceps or Ciaglia single-dilator techniques) for indications such as prolonged mechanical ventilation

SUMMARY:
The primary objective of this study was to determine the point prevalence of tracheostomy in adult intensive care units (ICUs) in Izmir and to evaluate indications, techniques, complications, timing, and short-term outcomes. This multicentre, descriptive point-prevalence study was conducted across seven adult ICUs on September 8, 2025. The study aimed to provide observational data on how tracheostomy is managed in a real-world clinical setting, focusing on the decision-making process and clinical characteristics associated with patient mortality

DETAILED DESCRIPTION:
This investigation was designed as a multicentre, descriptive point-prevalence study. On the specified prevalence day, all patients aged 18 years and older who had previously undergone tracheostomy using either surgical or percutaneous techniques in participating centers were included.

The data collection process involved:

* Documentation of ICU structural characteristics, including bed capacity and annual tracheostomy volumes.
* Systematic recording of patient demographics, comorbidities, tracheostomy indications, and the specific techniques used (e.g., Griggs guidewire dilating forceps, Ciaglia single-dilator, or surgical tracheostomy).
* Assessment of early and post-procedural complications.
* Evaluation of the time interval from endotracheal intubation to the tracheostomy procedure and identifying reasons for any delays.
* A 30-day follow-up to assess mortality outcomes for all included patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Hospitalized in the participating adult intensive care units on the point-prevalence day
* Previously undergone tracheostomy using either surgical or percutaneous techniques

Exclusion Criteria:

* Patients younger than 18 years
* Patients without a tracheostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients followed in seven different intensive care units in Izmir, Turkey, who required a tracheostomy for various clinical indications, primarily prolonged mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-09-08 (Actual); Primary Completion 2025-10-08 (Actual); Study Completion 2025-10-08 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30 days post-procedure
  The proportion of patients who died within 30 days following the tracheostomy procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir City Hospital, Izmir, Bayrakli, Turkey (Türkiye)